CLINICAL TRIAL: NCT00005754
Title: Coronary Artery Calcification in Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 97-661; R01HL061753 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Diabetes Mellitus; Diabetes Mellitus, Insulin-dependent
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To investigate the occurrence and associated risk factors for subclinical heart disease in persons with insulin-dependent diabetes mellitus (IDDM).

DETAILED DESCRIPTION:
BACKGROUND:

Approximately 10 percent of premature coronary artery disease (CAD) morbidity and mortality in the general population is due to insulin dependent diabetes mellitus (IDDM). By age 55, 35 percent of IDDM patents die of CAD, in contrast to only 8 percent of nondiabetic men and 4 percent of women. In the U.S., IDDM affects at least 750,000 persons and this number is growing rapidly as the effect of increasing incidence and improved survival. Tight blood glucose control can slow the development of microvascular complications but a protective effect on heart disease has not been convincingly demonstrated.

DESIGN NARRATIVE:

This observational population-based study evaluated cross- sectionally a population-based group of 656 IDDM patients aged 20-55 years and 764 of their non-diabetic spouse/partner controls using the electron-beam computed tomography (EBCT). Patients and controls were compared in terms of the amount and anatomical distribution of coronary artery calcium (CAC), a marker of atherosclerosis, and the left ventricular (LV) area, a marker of LV hypertrophy and diabetic cardiomyopathy. The demographic, metabolic, and behavioral factors associated with increased CACand LV area were defined. Standard epidemiological methods were used to determine the prevalence of clinical CAD, defined by previous MI, revascularization, or angina in the study population. In 100 asymptomatic high-risk IDDM patients (CAC greater than or equal to 20 or LV area greater than 60 cm2), in 50 low-risk patients (CAC and LV area below these cut-offs), and in 20 nondiabetic controls age-sex matched to the high-risk patients, ECG-gated rest-stress technetium-99m sestamibi single-photon emission computed tomographic imaging (MIBI SPECT) was performed. This helped to determine the presence of myocardial perfusion defects and to quantify myocardial perfusion reserve as well as to relate these findings anatomically to the distribution of CAC by EBCT. In addition, LV volumes, ejection fraction, wall motion and thickening were determined, and related to LV area by EBCT. Finally, the study cohort of 656 IDDM patients and 764 non diabetic spouses/partners were followed up for a period of 3 years to measure the change in CAC and LV area using a repeat EBCT and to identify the metabolic and behavioral risk factors for progression in these indices. Cause-specific mortality was monitored and all fatal and non-fatal cardiac events were ascertained. In the subgroup of 100 high-risk IDDM patients studied with the MIBI SPECT at the baseline and in all low-risk patients whose CAC increased by more than 50 during the follow-up, MIBI SPECT was used to evaluate the change in myocardial perfusion, LV volumes, ejection fraction, wall motion and thickening, as well as to relate these findings to the change in CAC and LV area by EBCT.

The study was extended to follow the cohort for an additional three years to achieve the following specific aims: 1. To determine, among type 1 diabetic (T1D) patients and comparable controls, the risk factors for: a. 6-year progression of electron-beam tomography (EBT) defined coronary calcification - marker of coronary atherosclerosis b. 6-year development of myocardial perfusion defects and changes in relative myocardial perfusion reserve defined using ECG-gated rest-stress technetium-99m MIBI SPECT imaging c. 6-year incidence of clinical CAD, defined by fatal and non-fatal MI, revascularization or angina, as well as stroke, peripheral artery disease and cause-specific mortality. 2. To develop a clinically useful measure of insulin sensitivity that is directly comparable between T1D patients and non-diabetic persons to more precisely determine the role of insulin resistance in development of premature CAC in type I diabetes.

ELIGIBILITY:
No eligibility criteria

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 656 IDDM patients aged 20-55 years and 764 of their non-diabetic spouse/partner controls
Sampling Method: Non-Probability Sample
Enrollment: 1420 (Actual)
Dates: Start 1999-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Progression of coronary artery calcification | 12 years

CONTACTS AND LOCATIONS:
Overall Officials: Marian Rewers, MD, PhD, Principal Investigator — University of Colorado, Denver

REFERENCES:
- [Background] Hokanson JE, Cheng S, Snell-Bergeon JK, Fijal BA, Grow MA, Hung C, Erlich HA, Ehrlich J, Eckel RH, Rewers M. A common promoter polymorphism in the hepatic lipase gene (LIPC-480C>T) is associated with an increase in coronary calcification in type 1 diabetes. Diabetes. 2002 Apr;51(4):1208-13. doi: 10.2337/diabetes.51.4.1208. PMID 11916946
- [Background] Wadwa RP, Kinney GL, Maahs DM, Snell-Bergeon J, Hokanson JE, Garg SK, Eckel RH, Rewers M. Awareness and treatment of dyslipidemia in young adults with type 1 diabetes. Diabetes Care. 2005 May;28(5):1051-6. doi: 10.2337/diacare.28.5.1051. PMID 15855566
- [Background] Maahs DM, Kinney GL, Wadwa P, Snell-Bergeon JK, Dabelea D, Hokanson J, Ehrlich J, Garg S, Eckel RH, Rewers MJ. Hypertension prevalence, awareness, treatment, and control in an adult type 1 diabetes population and a comparable general population. Diabetes Care. 2005 Feb;28(2):301-6. doi: 10.2337/diacare.28.2.301. PMID 15677783
- [Derived] Horton WB, Snell-Bergeon JK. Hemoglobin A1c Variability Metrics Predict Coronary Artery Calcium and Cardiovascular Events in Type 1 Diabetes: The CACTI Study. J Clin Endocrinol Metab. 2023 Jun 16;108(7):e444-e449. doi: 10.1210/clinem/dgad019. PMID 36637994
- [Derived] Basu A, Alman AC, Snell-Bergeon JK. Associations of Dietary Antioxidants with Glycated Hemoglobin and Insulin Sensitivity in Adults with and without Type 1 Diabetes. J Diabetes Res. 2022 Jun 25;2022:4747573. doi: 10.1155/2022/4747573. eCollection 2022. PMID 35789593
- [Derived] Basu A, Chien LC, Alman AC, Snell-Bergeon JK. Associations of dietary patterns and nutrients with coronary artery calcification and pericardial adiposity in a longitudinal study of adults with and without type 1 diabetes. Eur J Nutr. 2021 Oct;60(7):3911-3925. doi: 10.1007/s00394-021-02564-6. Epub 2021 Apr 27. PMID 33904996